CLINICAL TRIAL: NCT05686577
Title: Comment Diminuer Les hémocultures Inutiles : Construction et Validation d'un Score prédictif de positivité Des hémocultures en réanimation.
Brief Title: How to Reduce Unnecessary Blood Cultures: Construction and Validation of a Predictive Score for Blood Culture Positivity in Intensive Care
Acronym: PROBIty
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR200089 (PROBIty)
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Infection, Bacterial; Infection, Fungal; Bacteremia
Keywords: intensive care unit; blood culture; prediction; score
MeSH Terms: conditions — Bacterial Infections; Mycoses; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- learning database group: The results of blood cultures and the clinical elements of the patients in the first sample (1600 patients) will constitute the learning database. A supervised learning will be performed on these data in order to select a set of clinical elements allowing to define a predictive score of positive blood cultures
  Interventions: Other: no intervention
- validation database group: The score will be validated on the remaining sample (800 patients), independent of the first sample. Both samples will be constituted by randomization.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Prospective observational cohort consisting of all adult patients admitted to participating critical care units (ICU and CCU) during the study period, with blood cultures collected as part of their care, and who did not express any objection to participating.

For each patient, data will be collected prospectively for each blood culture set collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older
* Patient admitted to an ICU or ICU
* patient with a blood culture sample as part of care

Exclusion Criteria:

* Patient already included in this study during a previous hospitalisation
* Opposition expressed for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critical care patient with suspected infection.
Sampling Method: Non-Probability Sample
Enrollment: 2411 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Area under the ROC curve of the predictive performance of the score for predicting bacteremia or fungemia. | day 1- day 28

SECONDARY OUTCOMES:
Area under the ROC curve of the diagnostic performance of body temperature to predict bacteremia or fungemia; | day 1- day 28
Area under the ROC curve of the diagnostic performance of the Shapiro score for predicting bacteremia or fungemia; | day 1- day 28
Proportion of bacteremia or fungemia identified by blood cultures in patients on antibiotic therapy and broad-spectrum antibiotic therapy, and factors associated with these bacteremias or fungemias; | day 1- day 28
Comparison of the diagnostic performance of the score in predicting bacteremia or fungemia observed during the first 48 hours of hospitalization to later bacteremias; | 48 hours
Descriptive study of the contribution of blood cultures, whatever their results, to the prescription of anti-infectives. | day 1- day 28
Efficiency of the new predictive score for blood culture positivity in Intensive Care, as compared with body temperature and Shapiro score, measured by two Incremental Cost-Effectiveness Ratios (ICER): ICER (incremental cost per additional well-detecte | less than 1 month
  A tree decision model will compare three strategies for predicting positive blood cultures: the new predictive score, body temperature and Shapiro score. Within-trial data will be used to define the model parameters. The model will consider the costs related to the implementation of the strategies, blood cultures, and potential delays in patient management. This will result in the estimation of the two ICERs.

CONTACTS AND LOCATIONS:
Overall Officials: Denis GAROT, Principal Investigator — University Hospital, Tours
Locations (10):
- France (10):
  - CHU Brest, Brest
  - CHU Dijon, Dijon
  - CHD La Roche sur Yon, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CHU Nantes, Nantes
  - CHR Orléans, Orléans
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHIU Strasbourg, Strasbourg
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335
- [Background] Rhee C, Dantes R, Epstein L, Murphy DJ, Seymour CW, Iwashyna TJ, Kadri SS, Angus DC, Danner RL, Fiore AE, Jernigan JA, Martin GS, Septimus E, Warren DK, Karcz A, Chan C, Menchaca JT, Wang R, Gruber S, Klompas M; CDC Prevention Epicenter Program. Incidence and Trends of Sepsis in US Hospitals Using Clinical vs Claims Data, 2009-2014. JAMA. 2017 Oct 3;318(13):1241-1249. doi: 10.1001/jama.2017.13836. PMID 28903154
- [Background] Goto M, Al-Hasan MN. Overall burden of bloodstream infection and nosocomial bloodstream infection in North America and Europe. Clin Microbiol Infect. 2013 Jun;19(6):501-9. doi: 10.1111/1469-0691.12195. Epub 2013 Mar 8. PMID 23473333
- [Background] McNamara JF, Righi E, Wright H, Hartel GF, Harris PNA, Paterson DL. Long-term morbidity and mortality following bloodstream infection: A systematic literature review. J Infect. 2018 Jul;77(1):1-8. doi: 10.1016/j.jinf.2018.03.005. Epub 2018 May 7. PMID 29746948
- [Background] Patel R. New Developments in Clinical Bacteriology Laboratories. Mayo Clin Proc. 2016 Oct;91(10):1448-1459. doi: 10.1016/j.mayocp.2016.06.020. Epub 2016 Aug 21. PMID 27552910
- [Background] Leyssene D, Gardes S, Vilquin P, Flandrois JP, Carret G, Lamy B. Species-driven interpretation guidelines in case of a single-sampling strategy for blood culture. Eur J Clin Microbiol Infect Dis. 2011 Dec;30(12):1537-41. doi: 10.1007/s10096-011-1257-3. Epub 2011 Apr 18. PMID 21499970
- [Background] Dargere S, Cormier H, Verdon R. Contaminants in blood cultures: importance, implications, interpretation and prevention. Clin Microbiol Infect. 2018 Sep;24(9):964-969. doi: 10.1016/j.cmi.2018.03.030. Epub 2018 Apr 3. PMID 29621616
- [Background] Kirn TJ, Weinstein MP. Update on blood cultures: how to obtain, process, report, and interpret. Clin Microbiol Infect. 2013 Jun;19(6):513-20. doi: 10.1111/1469-0691.12180. Epub 2013 Mar 13. PMID 23490046
- [Background] Opota O, Croxatto A, Prod'hom G, Greub G. Blood culture-based diagnosis of bacteraemia: state of the art. Clin Microbiol Infect. 2015 Apr;21(4):313-22. doi: 10.1016/j.cmi.2015.01.003. Epub 2015 Jan 16. PMID 25753137
- [Background] Lamy B, Dargere S, Arendrup MC, Parienti JJ, Tattevin P. How to Optimize the Use of Blood Cultures for the Diagnosis of Bloodstream Infections? A State-of-the Art. Front Microbiol. 2016 May 12;7:697. doi: 10.3389/fmicb.2016.00697. eCollection 2016. PMID 27242721
- [Background] Lin HH, Liu YF, Tien N, Ho CM, Hsu LN, Lu JJ. Evaluation of the blood volume effect on the diagnosis of bacteremia in automated blood culture systems. J Microbiol Immunol Infect. 2013 Feb;46(1):48-52. doi: 10.1016/j.jmii.2012.03.012. Epub 2012 Jun 26. PMID 22738875
- [Background] Snyder SR, Favoretto AM, Baetz RA, Derzon JH, Madison BM, Mass D, Shaw CS, Layfield CD, Christenson RH, Liebow EB. Effectiveness of practices to reduce blood culture contamination: a Laboratory Medicine Best Practices systematic review and meta-analysis. Clin Biochem. 2012 Sep;45(13-14):999-1011. doi: 10.1016/j.clinbiochem.2012.06.007. Epub 2012 Jun 16. PMID 22709932
- [Background] Caldeira D, David C, Sampaio C. Skin antiseptics in venous puncture-site disinfection for prevention of blood culture contamination: systematic review with meta-analysis. J Hosp Infect. 2011 Mar;77(3):223-32. doi: 10.1016/j.jhin.2010.10.015. Epub 2010 Dec 30. PMID 21194791
- [Background] Dargere S, Parienti JJ, Roupie E, Gancel PE, Wiel E, Smaiti N, Loiez C, Joly LM, Lemee L, Pestel-Caron M, du Cheyron D, Verdon R, Leclercq R, Cattoir V; UBC study group. Unique blood culture for diagnosis of bloodstream infections in emergency departments: a prospective multicentre study. Clin Microbiol Infect. 2014 Nov;20(11):O920-7. doi: 10.1111/1469-0691.12656. Epub 2014 Jun 14. PMID 24766148
- [Background] Cockerill FR 3rd, Hughes JG, Vetter EA, Mueller RA, Weaver AL, Ilstrup DM, Rosenblatt JE, Wilson WR. Analysis of 281,797 consecutive blood cultures performed over an eight-year period: trends in microorganisms isolated and the value of anaerobic culture of blood. Clin Infect Dis. 1997 Mar;24(3):403-18. doi: 10.1093/clinids/24.3.403. PMID 9114192
- [Background] Andrews AL, Simpson AN, Heine D, Teufel RJ 2nd. A Cost-Effectiveness Analysis of Obtaining Blood Cultures in Children Hospitalized for Community-Acquired Pneumonia. J Pediatr. 2015 Dec;167(6):1280-6. doi: 10.1016/j.jpeds.2015.09.025. Epub 2015 Oct 9. PMID 26456740
- [Background] Coburn B, Morris AM, Tomlinson G, Detsky AS. Does this adult patient with suspected bacteremia require blood cultures? JAMA. 2012 Aug 1;308(5):502-11. doi: 10.1001/jama.2012.8262. PMID 22851117
- [Background] Yamamoto S, Yamazaki S, Shimizu T, Takeshima T, Fukuma S, Yamamoto Y, Tochitani K, Tsuchido Y, Shinohara K, Fukuhara S. Body Temperature at the Emergency Department as a Predictor of Mortality in Patients With Bacterial Infection. Medicine (Baltimore). 2016 May;95(21):e3628. doi: 10.1097/MD.0000000000003628. PMID 27227924
- [Background] Eliakim-Raz N, Bates DW, Leibovici L. Predicting bacteraemia in validated models--a systematic review. Clin Microbiol Infect. 2015 Apr;21(4):295-301. doi: 10.1016/j.cmi.2015.01.023. Epub 2015 Feb 10. PMID 25677625
- [Background] Shapiro NI, Wolfe RE, Wright SB, Moore R, Bates DW. Who needs a blood culture? A prospectively derived and validated prediction rule. J Emerg Med. 2008 Oct;35(3):255-64. doi: 10.1016/j.jemermed.2008.04.001. Epub 2008 May 16. PMID 18486413
- [Background] Laukemann S, Kasper N, Kulkarni P, Steiner D, Rast AC, Kutz A, Felder S, Haubitz S, Faessler L, Huber A, Fux CA, Mueller B, Schuetz P. Can We Reduce Negative Blood Cultures With Clinical Scores and Blood Markers? Results From an Observational Cohort Study. Medicine (Baltimore). 2015 Dec;94(49):e2264. doi: 10.1097/MD.0000000000002264. PMID 26656373
- [Background] Peres Bota D, Melot C, Lopes Ferreira F, Vincent JL. Infection Probability Score (IPS): A method to help assess the probability of infection in critically ill patients. Crit Care Med. 2003 Nov;31(11):2579-84. doi: 10.1097/01.CCM.0000094223.92746.56. PMID 14605527
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Hanley JA, McNeil BJ. The meaning and use of the area under a receiver operating characteristic (ROC) curve. Radiology. 1982 Apr;143(1):29-36. doi: 10.1148/radiology.143.1.7063747.